CLINICAL TRIAL: NCT05813262
Title: Patient Opinions Regarding General Anesthesia, Before and After Having Undergone a Procedure.
Status: Completed | Type: Observational
Sponsor: Alabama College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Dr. Gordon MacGregor, Associate Professor of Pharmacology, Alabama College of Osteopathic Medicine
Other Study IDs: HS220404
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia
Keywords: General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this survey will be to assess the opinions and reticence of patients who have undergone surgical procedures that required the usage of general anesthesia both before they underwent the procedure and afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Have experience with general anesthesia.

Exclusion Criteria:

* Anyone who has not undergone a procedure using general anesthesia and who will not undergo such a procedure within the next 6 months.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from physicians offices in Alabama and Florida. Recruitment will be via posters displayed at one of these three locations. Participants will also be recruited via social media platforms.
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Perceived level of anxiety towards general anesthesia | From exposure to general anesthesia until survey completion by September 2022
  The perceived level of anxiety (on a scale of 1 to 10) before and after undergoing general anesthesia
Perceived level of danger towards general anesthesia | From exposure to general anesthesia until survey completion by September 2022
  The perceived level of danger (on a scale of 1 to 10) before and after undergoing general anesthesia
Perceived side effects of general anesthesia | From exposure to general anesthesia until survey completion by September 2022
  Description of perceived side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Ashford Clinic, Ashford, Alabama, United States

IPD SHARING:
Plan to Share IPD: No